CLINICAL TRIAL: NCT01440738
Title: Effectiveness of a Group Intervention to Promote Health Through a Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI09/90746
Record Dates: First submitted 2010-06-21; First posted 2011-09-26 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2011-09

CONDITIONS: Healthy
Keywords: general population

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- health workshops (Experimental): Health promotion group intervention
  Interventions: Behavioral: health workshops
- comparison group (No Intervention): usual care

INTERVENTIONS:
Behavioral: health workshops — health workshops in relation to: Increase knowledge of healthy habits (physical activity, diet), incorporate and maintain a balanced diet. Incorporate and maintain regular physical activity
  Arms: health workshops

SUMMARY:
Objectives

Main objective: Assessing the effectiveness of the health workshops, in terms of quality of life.

Secondary: To determine the effectiveness of the health workshops in relation to: Increase knowledge of healthy habits (physical activity, diet), incorporate and maintain a balanced diet. Incorporate and maintain regular physical activity; Keep variables related to risk factors (BP, Weight, Cholesterol) within normal limits, reduce cardiovascular risk (RCV). To estimate costs.

Methodology

Design: randomized controlled trial comparing a group of patients who performed the health workshops with a control group with similar characteristics.

Scope of the Study: The study was conducted in 54 health centers of Barcelona city.

Subjects of study: general population between 18 and 65 years who consent to. 188 people with speech (have conducted workshops for health) and 188 people without (not made health workshops. Data Analysis: T- test to compare the differences between quantitative variables or equivalent non-parametric if the distribution of the variable does not meet criteria of normality (Kolmogorov-Smirnov).

DETAILED DESCRIPTION:
This is the evaluation of an educational activity to promote health in the general population in order to establish healthy habits and changes in quality of life.

We have designed a proposal for a workshop aimed at general public health which includes biological, psychological, social, cultural and spiritual health related and welfare. It is structured in 12 sessions that will provide tools that facilitate the involvement of people in maintaining their health.

Content of the sessions: Breathing and Snuff. Food. Disposal. Physical activity. Sleep and rest. Appropriate clothing. Hygiene. Avoid danger. Communicate feelings and emotions. Feel useful. Recreational activities. Each participant is given a folder and at the end of each session a summary sheet of the same with the aim that at the end of the course have a reference material.

To validate this material is piloted with the participation of 13 persons. Participants completed the SF36 questionnaire at the beginning and end of the workshop.

ELIGIBILITY:
Inclusion Criteria:

* General population between 18 and 65 years who consent to participate.

Exclusion Criteria:

* Difficulty to maintain their participation for 12 months.
* Difficult to understand and speak Catalan or Spanish language.
* Severe mental health problems.
* Other health problems that their participation was not appropriate or fail to follow up planned (terminally ill, serious organic disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of life | 0, 3, 6 and 12 months
  Health Ralated Quality of Life (EuroQol 5D-3L)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonia Campo Osaba, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Institut català de la salut, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Campo Osaba MA, Del Val JL, Lapena C, Laguna V, Garcia A, Lozano O, Martin Z, Rodriguez R, Borras E, Orfila F, Tierno MT. The effectiveness of a health promotion with group intervention by clinical trial. Study protocol. BMC Public Health. 2012 Mar 19;12:209. doi: 10.1186/1471-2458-12-209. PMID 22429693
- See also: Related Info — https://doi.org/10.1186/1471-2458-12-209